CLINICAL TRIAL: NCT06537141
Title: Role of Selective Embolization of Thyroid Arteries (SETA) as an Adjunctive or Definitive Treatment for Different Thyroid Disorders
Brief Title: Role of Embolization of Thyroid Arteries as a Treatment for Different Thyroid Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abdelRahman Ahmad abdAllah, assistant lecturer, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3ekremaH
Record Dates: First submitted 2024-07-12; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Graves Disease; Goiter, Nodular; Goiter Malignant; Goiter Diffuse
Keywords: Embolization of thyroid arteries
MeSH Terms: conditions — Graves Disease; Goiter, Nodular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- graves disease patients (Active Comparator)
  Interventions: Procedure: selective embolization of thyroid arteries (SETA)
- multinodular goiter (Active Comparator)
  Interventions: Procedure: selective embolization of thyroid arteries (SETA)

INTERVENTIONS:
Procedure: selective embolization of thyroid arteries (SETA) — selective embolization of thyroid arteries

SUMMARY:
To investigate the safety and efficacy of selective embolization of thyroid arteries (SETA) as adjunctive or definitive treatment in different thyroid disorders

DETAILED DESCRIPTION:
In graves disease Traditional forms of treatment of the thyroid diseases: pharmacotherapy, radioiodine therapy and surgery can not always be applied. Intolerance, side effects of antithyroid drugs, low iodine uptake, high risk of surgery or disagreement with the proposed treatment was the reason for seeking alternative treatment methods.

Also in cases of large sized thyroid nodule and retrosternal extension, surgery may carries out a lot of comorbidities .

With the development of interventional radiology, and gained experience in the use of arterial embolization, this method has become possible to use in treatment of thyroid diseases. The essence of this treatment is to shut down blood flow in major arteries of the thyroid by direct injection of embolizing materials (PVA) into the vessel's.

. The consequence of acute ischemia is necrosis of the glandular tissue in a field being supplied by this artery. Further repair processes and fibrosis lead to a reduction of active thyroid hormone synthesis and restriction of thyroid gland. Effects of embolization on angiogenesis, apoptosis and autoimmune reactions contribute to compensation thyroid function and significant reduction a goiter volume in course of Graves' disease. Preoperative selective embolization of a huge goiter or thyroid cancer improves surgery outcomes, reduces the risk of hemorrhage and damage to surrounding tissue. Palliative use of embolization in advanced stages of thyroid cancer reduces symptoms and improves quality of life. Little invasive nature of this procedure, the lack of serious undesirable coincidence makes embolization of thyroid arteries an attractive form of a therapy, which may become a therapeutic option in many difficult clinical situations and improve the clinical effectiveness of treatment of thyroid disease

ELIGIBILITY:
Inclusion Criteria:

A- diffuse and Nodular goiter:

B-Toxic goiter:

C-Thyroid cancer:

Exclusion Criteria:

A. Significant bleeding diathesis. B. Contraindication for contrast media (renal impairment or allergy). C. Severe atherosclerotic disease prevent arterial catheterization. D. Refusal of signing a consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety of selective embolization of thyroid arteries (SETA) as adjunctive or definitive treatment in different thyroid disorders | Up to 12 months follow up after embolization
  Safety measured according to incidence of major and minor complications compared to thyroidectomy.
To investigate the efficacy of selective embolization of thyroid arteries (SETA) as adjunctive or definitive treatment in different thyroid disorders | Up to 12 months follow up after embolization
  in hyperfunctiong (toxic) disorders Efficacy measured according to thyroid profile levels in certain time interval post procedure, every 3 months time interval and rate of hyper functioning recurrence in comparison to thyroidectomy.
  In diffuse or nodular goiter we measure efficacy by percentage of size reduction post procedure in comparison to primary size just before procedure